CLINICAL TRIAL: NCT01406041
Title: Disturbance of Water and Sodium Metabolism After Surgery of Sellar Lesions, and Correspond Clinical Strategy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Pan Jun, department of neurosurgery, Southern Medical University, China
Other Study IDs: The department of Neurosurgery
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: The Patients Suffered With Sellar Diseases; The Fluid and Electrolyte Imbalance Happened After Surgery
Keywords: Fluid and electrolyte imbalance; Hyponatremia; Hypernatremia; Electrolytes disorder
MeSH Terms: conditions — Hyponatremia; Hypernatremia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diseases: 1. Pituitary adenomas; 2. Craniopharyngioma; 3. Sellar germinoma; 4. Sellar tuberalis meningioma; 5. Hypophystis; 6. Sellar glioma; 7. Rathke's cleft cyst; 8. Hypothalamic hamartoma
  Interventions: Biological: Chemical and physical detection

INTERVENTIONS:
Biological: Chemical and physical detection — CVP, Urine volume per day, Blood electrolytes, Urine sodium per day, Pituitrin

SUMMARY:
The fluid and electrolyte imbalance (FEI) is pretty common encountered during the clinical process of patients suffered sellar lesions. Moreover, if the patients are undergone the surgery for remove the lesion, FEI happens in all cases without exception. Hypo- and hyper-natremia is the most common electrolyte disorder, which is directly correlated to the patients' outcome. However, in clinical works, different sellar diseases cause variant features of FEI. For example, after the surgery of craniopharyngioma, the hyponatremia and hypernatremia always happen alternatively even without any precursor manifestation. Under this situation, it is quite difficult for fluid supplement. In contrast, the severe FEI will cause poor outcome, even death. So it is necessary to systematically collect and review the clinical data of sellar lesions. Through the analysis of variant FEI patterns of sellar diseases, more precise strategy for clinical fluid replacement will be proposed.

ELIGIBILITY:
Inclusion Criteria:

* 1. Suffered with sellar disease
* 2. Udergone surgery
* 3. Have sufficient presurgical and postsurgical clinical data (Including MRI, CT, physical and chemical detection results)

Exclusion Criteria:

* 1. Without sufficitent clincal data
* 2. No surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presented in our department suffered with sellar diseases
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2011-02; Primary Completion 2020-01-30 (Actual); Study Completion 2021-05-12 (Estimated)

PRIMARY OUTCOMES:
Blood sodium | 24 hours
  Normal: 135~155

SECONDARY OUTCOMES:
Urine sodium | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- The department of Neurosurgery, Nanfang hospital, Guangzhou, Guangdong, China